CLINICAL TRIAL: NCT05840497
Title: Efecto Del Ejercicio De Fuerza-resistencia En La Disminución De La Diabetes Gestacional En Gestantes Con Sobrepeso U Obesidad
Brief Title: Effect of Strength-resistance Exercise in the Reduction of Gestational Diabetes in Pregnant Women with Overweight or Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Principal Investigator, Olga Sanz, MD, Fundacion Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI_2022/126
Record Dates: First submitted 2023-04-13; First posted 2023-05-03 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Diabetes, Gestational
Keywords: Exercise; Weight gain; Pregnant; Obese; Overweight
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity; Weight Gain; Obesity; Overweight | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistance exercise (Experimental)
  Interventions: Other: Resistance exercise
- Control Group (No Intervention): Standard control and usual recommendations.

INTERVENTIONS:
Other: Resistance exercise — The intervention group will train 3 times per week (30 minutes with 15 min warm-up). The resistance exercise is described as the voluntary contraction of the skeletal muscle of a particular muscle group against some type of resistance, using light weights, elastic bands or the weight of the body itself.
  Patients will be offered online sessions, they will receive a document with recommendations and a link to the videos with instructions.
  .
  Arms: Resistance exercise

SUMMARY:
The aim of this trial is to test the efficacy of regular resistance exercise in early pregnancy to prevent gestational diabetes mellitus in overweight/ obese pregnant women.

DETAILED DESCRIPTION:
The growing rate of obesity is a major public health problem in the West, where 28% of pregnant women are overweight and 11% are obese. Worldwide, 50% of pregnant women are obese or overweight.

One of the problems directly related to obesity is gestational diabetes. In fact, its prevalence is increasing as the prevalence of obesity increases, as well as other complications of pregnancy. The prevalence of gestational diabetes in our environment is 6-12%.

Compared with pregnant women with BMI <25 kg/m2, pregnancies among women with obesity are at increased risk of several adverse outcomes, including early pregnancy loss, congenital anomalies, stillbirth, pregnancy-associated hypertension, preterm birth and postterm, gestational diabetes mellitus, multiple gestation, cesarean delivery, and birth of a macrosome.

The consequences of obesity in pregnant women can be decreased through physical activity. This hypothesis is due to several mechanisms: reduction of blood pressure, improvement of the lipid profile, reduction of oxidative stress and the proinflammatory state.

In recent years, scientific societies have published new recommendations on physical exercise in pregnant women with clear guidelines. Even this, less than 15% of patients do the recommended exercise. Usually the recommended exercise is aerobic and in the group of obese and overweight patients this type of exercise requires more effort and time, with the consequent worse adherence.

In non-pregnant patients, exercise has been shown to be related to a decrease in cardiovascular risk and DM2. However, in pregnant patients, a meta-review of systematic reviews has shown that although lifestyle interventions decrease weight gain, they do not have a clear benefit in terms of maternal-fetal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥25 kg/m2
* Singleton pregnancies

Exclusion Criteria:

* Chronic hypertension
* Pre-pregnancy DM (type I or 2 diabetes mellitus)
* Cardiovascular disease
* History of preterm delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Gestational diabetes | 24-28 gestational weeks
  Gestational diabetes mellitus (GDM) is defined as any degree of glucose intolerance with onset or first recognition during pregnancy:
  * O'Sullivan Test: if this is pathological;
  * SOG with 100 gr of glucose (GDM is diagnosed when 2 or more altered values: basal glycemia >105 mg / dl, at 1 hour >190 mg / dl, at 2h glycemia >165 mg / dl, at 3h glycemia >145 gr/dl).

SECONDARY OUTCOMES:
Weight gain and excessive body weight gain | From baseline visit to the third trimester visit
  Determined by IOM (Institute of Medicine) guideline
Maternal and fetal pregnancy outcomes | At birth
  Newborn weight, preterm deliveries, Apgar score and pH of umbilical cord, duration of labour and delivery mode

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Miguel Servet/Navarrabiomed, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhattacharya S, Campbell DM, Liston WA, Bhattacharya S. Effect of Body Mass Index on pregnancy outcomes in nulliparous women delivering singleton babies. BMC Public Health. 2007 Jul 24;7:168. doi: 10.1186/1471-2458-7-168. PMID 17650297
- [Background] Xu MY, Guo YJ, Zhang LJ, Lu QB. Effect of individualized weight management intervention on excessive gestational weight gain and perinatal outcomes: a randomized controlled trial. PeerJ. 2022 Mar 8;10:e13067. doi: 10.7717/peerj.13067. eCollection 2022. PMID 35282280
- [Background] Roberts JM, Bodnar LM, Patrick TE, Powers RW. The Role of Obesity in Preeclampsia. Pregnancy Hypertens. 2011 Jan 1;1(1):6-16. doi: 10.1016/j.preghy.2010.10.013. PMID 21532964
- [Background] Domingues MR, Bassani DG, da Silva SG, Coll Cde V, da Silva BG, Hallal PC. Physical activity during pregnancy and maternal-child health (PAMELA): study protocol for a randomized controlled trial. Trials. 2015 May 24;16:227. doi: 10.1186/s13063-015-0749-3. PMID 26003406
- [Background] Fair F, Soltani H. A meta-review of systematic reviews of lifestyle interventions for reducing gestational weight gain in women with overweight or obesity. Obes Rev. 2021 May;22(5):e13199. doi: 10.1111/obr.13199. Epub 2021 Jan 18. PMID 33459493
- [Background] Magro-Malosso ER, Saccone G, Di Mascio D, Di Tommaso M, Berghella V. Exercise during pregnancy and risk of preterm birth in overweight and obese women: a systematic review and meta-analysis of randomized controlled trials. Acta Obstet Gynecol Scand. 2017 Mar;96(3):263-273. doi: 10.1111/aogs.13087. PMID 28029178
- [Background] Petrov Fieril K, Glantz A, Fagevik Olsen M. The efficacy of moderate-to-vigorous resistance exercise during pregnancy: a randomized controlled trial. Acta Obstet Gynecol Scand. 2015 Jan;94(1):35-42. doi: 10.1111/aogs.12525. Epub 2014 Nov 13. PMID 25287282
- [Background] Barakat R, Ruiz JR, Stirling JR, Zakynthinaki M, Lucia A. Type of delivery is not affected by light resistance and toning exercise training during pregnancy: a randomized controlled trial. Am J Obstet Gynecol. 2009 Dec;201(6):590.e1-6. doi: 10.1016/j.ajog.2009.06.004. Epub 2009 Jul 15. PMID 19608151
- [Background] Xie Y, Zhao H, Zhao M, Huang H, Liu C, Huang F, Wu J. Effects of resistance exercise on blood glucose level and pregnancy outcome in patients with gestational diabetes mellitus: a randomized controlled trial. BMJ Open Diabetes Res Care. 2022 Apr;10(2):e002622. doi: 10.1136/bmjdrc-2021-002622. PMID 35383101
- [Background] Wang C, Wei Y, Zhang X, Zhang Y, Xu Q, Sun Y, Su S, Zhang L, Liu C, Feng Y, Shou C, Guelfi KJ, Newnham JP, Yang H. A randomized clinical trial of exercise during pregnancy to prevent gestational diabetes mellitus and improve pregnancy outcome in overweight and obese pregnant women. Am J Obstet Gynecol. 2017 Apr;216(4):340-351. doi: 10.1016/j.ajog.2017.01.037. Epub 2017 Feb 1. PMID 28161306